CLINICAL TRIAL: NCT06654817
Title: Evaluation of Combination Therapy with Ofatumumab and Systemic Corticosteroids for Pemphigus: a Multi-center Cohort Study
Brief Title: Efficacy and Safety Evaluation of Anti-CD20 Monoclonal Antibody Combined with Azathioprine and Corticosteroids in the Treatment of Pemphigus Vulgaris
Status: Completed | Type: Observational
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, Clinical Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH OfFMU|2024]565
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pemphigus; Pemphigus Vulgaris (PV)
Keywords: Pemphigus
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- experimental group: ofatumumab combined with corticosteroids versus corticosteroids
  To compare the efficacy and safety of two treatment strategies: ofatumumab combined with corticosteroids versus corticosteroids along with azathioprine, in pemphigus patients.
  A prospective cohort study was conducted, following patients for 36 weeks from January 1, 2023, to April 30, 2024. Patients meeting the diagnostic criteria were nonrandomly grouped based on screening results. The primary endpoints were time to disease control and skin healing. Secondary endpoints included complete remission rates, relapse rates, corticosteroid doses, pemphigus disease area index (PDAI), dermatology life quality index (DLQI), visual analogue scale (VAS) pain scores, CD19+ B cell percentages, desmoglein-specific antibodies, and adverse events.
  Interventions: Drug: Ofatumumab subcutaneous injection
- control group: the standard treatment of corticosteroids plus azathioprine

INTERVENTIONS:
Drug: Ofatumumab subcutaneous injection — To compare the efficacy and safety of two treatment strategies: ofatumumab combined with corticosteroids versus corticosteroids along with azathioprine, in pemphigus patients.
  Groups: experimental group

SUMMARY:
A prospective cohort study was conducted, following patients for 36 weeks from January 1, 2023, to April 30, 2024. Patients meeting the diagnostic criteria were nonrandomly grouped based on screening results. The primary endpoints were time to disease control and skin healing. Secondary endpoints included complete remission rates, relapse rates, corticosteroid doses, pemphigus disease area index (PDAI), dermatology life quality index (DLQI), visual analogue scale (VAS) pain scores, CD19+ B cell percentages, desmoglein-specific antibodies, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

- Patients with moderate to severe pemphigus who have poor control of previous external medications and require systemic treatment have a PDAI (Pemphigus Area and Activity Score) greater than 9 points.

Exclusion Criteria:

* Patients with serious basic diseases, with hepatitis B and three positive cases, and with a history of immunoglobulin related diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with alopecia areata
  Inclusion Criteria:
  Patients with moderate to severe pemphigus who have poor control of previous external medications and require systemic treatment have a PDAI (Pemphigus Area and Activity Score) greater than 9 points.
  Exclusion Criteria:
  * Patients with serious basic diseases, with hepatitis B and three positive cases, and with a history of immunoglobulin related diseases.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Pemphigus Disease Area Index (PDAI） | 36 week
  Pemphigus Disease Area Index (PDAI). PDAI activity score cutoffs were defined as 0 to 8 for mild, 9 to 24 for moderate, and 25 or higher for severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Zheyu Zheyu Zhuang, Study Director — Chao Ji
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided